CLINICAL TRIAL: NCT01019291
Title: Aldehyde and Nitrogen Dioxide at Homes: Measurement of the Exposure and Their Role on Allergic Asthma
Brief Title: Role of Indoor Pollutants on House Dust Mite Allergic Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Directeur de la Recherche Clinique et des Innovations, Hôpitaux Universitaires de Strasbourg
Allocation: Randomized | Masking: Double
Other Study IDs: 3965
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Asthma; Allergy to House Dust Mite
Keywords: Indoor pollutants
MeSH Terms: conditions — Dust Mite Allergy | interventions — Formaldehyde

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NO2 (Experimental): NO2 400 µg/m3
  Interventions: Other: Formaldehyde and NO2 (Exposure to indoor pollutants)
- Formaldehyde (Experimental): Formaldehyde 100 µg/m3
  Interventions: Other: Formaldehyde and NO2 (Exposure to indoor pollutants)
- NO2 + Formaldehyde (Experimental): mixture of Formaldehyde and NO2
  Interventions: Other: Formaldehyde and NO2 (Exposure to indoor pollutants)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (Exposure to indoor pollutants)

INTERVENTIONS:
Other: Formaldehyde and NO2 (Exposure to indoor pollutants) — Exposure to indoor pollutants (Formaldehyde and NO2) in a randomized way, followed by bronchial challenge test with house dust mite extract.
  Arms: Formaldehyde; NO2; NO2 + Formaldehyde
Other: Placebo (Exposure to indoor pollutants) — Exposure to indoor pollutants (placebo) in a randomized way, followed by bronchial challenge test with house dust mite extract.
  Arms: Placebo

SUMMARY:
It seems that the aldehydes and NO2, at the levels found indoor, could be the aggravating factors for an allergic response. However this effect has not been demonstrated. The investigators plan to study the effect of exposure to standard doses of these pollutants on the bronchial reactivity as measured by bronchial challenge tests with dust mite extract in volunteers asthmatic, allergic to house dust mite.

ELIGIBILITY:
Inclusion criteria:

* M/F 18-50 years of age
* History of intermittent HDM allergic asthma-FEV1 > 80%
* Non smokers or smokers with smoking < 10 PY

Exclusion criteria:

* Persistent asthma and FEV1<80%
* Allergic to pets and pets at home

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DE BLAY, MD, Principal Investigator — Service de Pneumologie, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg
Locations (1):
- Unité de Pneumologie, d'Allergologie et de Pathologie Respiratoire de l'Environnement, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France